CLINICAL TRIAL: NCT01231152
Title: The Relation of Obesity With Metabolic Disorders, Inflammation Markers and Arterial Blood Pressure With Preclinical Target-organ Damage in Children and Young Adolescents.
Brief Title: The Impact of Obesity on Children and Adolescents.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, George S. Stergiou, Associate Professor of Medicine and Hypertension, University of Athens
Other Study IDs: OB10
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-05

CONDITIONS: Obesity; Cardiovascular Risk Factors
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to investigate the association of obesity with arterial blood pressure, atherosclerosis, target organ damage (heart, arteries, kidney) and insulin resistance in children and young adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (85th<BMI<95th percentile) and obese (BMI>=95th percentile) children and adolescents
* No medication treatment (apart from bronchodilators, T4 in euthyroid children)
* No severe mental problem
* Parents' and patients' signed consent

Exclusion Criteria:

* Severe chronic or acute cardiac disease or other severe chronic or acute disease
* Any acute inflammation
* Familial dyslipidemia
* Clinical hypothyroidism or other endocrinopathy
* Poor compliance.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents referred for increased body weight.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure levels, Target organ damage (Left Ventricular Hypertrophy, IMT, pulse wave velocity, microalbuminuria), Insulin Resistance | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George S Stergiou, Principal Investigator — University of Athens
Locations (1):
- Hypertension Center, Third Department of Medicine, University of Athens, Athens, Greece